CLINICAL TRIAL: NCT04810117
Title: Monitoring the Patterns of IgG/IgM Antibodies in Asymptomatic/Symptomatic COVID-19 Patients
Brief Title: Monitoring the IgG/IgM Antibodies in COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: University of Sargodha (Other)
Collaborators: Shanghai Jiao Tong University School of Biomedical engineering (Unknown)
Responsible Party: Principal Investigator, Muhammad Fayyaz ur Rehman, Lecturer, University of Sargodha
Other Study IDs: 15032021-1
Record Dates: First submitted 2021-03-19; First posted 2021-03-22 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: COVID-19 Infections
Keywords: COVID-19; SARS-CoV-2; Humoral response
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (6):
- COVID-19 PCR positive patients who are not yet vaccinated: Patients test positive with PCR and recovered from COVID-19
  Interventions: Diagnostic Test: Serodiagnosis of IgG and IgM
- COVID-19 patients with obvious symptoms who are not yet vaccinated: COVID-19 patients with obvious symptoms but PCR test was not conducted for them
  Interventions: Diagnostic Test: Serodiagnosis of IgG and IgM
- COVID-19 suspected patients with no symptoms who are not yet vaccinated: COVID-19 suspected patients with no symptoms but came in obvious contact with infected environmental/biological samples
  Interventions: Diagnostic Test: Serodiagnosis of IgG and IgM
- COVID-19 PCR positive patients who are vaccinated: COVID-19 suspected patients who have got either one or two doses of vaccine
  Interventions: Diagnostic Test: Serodiagnosis of IgG and IgM
- Healthy Individuals who are vaccinated: Control group
  Interventions: Diagnostic Test: Serodiagnosis of IgG and IgM
- Healthy Individuals who are not vaccinated: Control group
  Interventions: Diagnostic Test: Serodiagnosis of IgG and IgM

INTERVENTIONS:
Diagnostic Test: Serodiagnosis of IgG and IgM — IgG and IgM antibodies will be detected in COVID-19 patients

SUMMARY:
The COVID-19 was declared a global pandemic by WHO more than a year ago, and the world is still experiencing a state of global emergency. This disease is caused by a novel RNA coronavirus suspected to originate in animals like bats and pangolin. Coronaviruses found in humans can be divided into seven classes, and out of them, three, i.e., MERS-CoV, SARS-CoV, and SARS-CoV-2, lead to global outbreaks. SARS-CoV-2 has claimed more than 120 million confirmed global cases of the COVID-19, where more than 26 million fatalities have also been recorded by the mid of March 2021. Many drugs have been repurposed and employed, but no specific antiviral medicine has been approved by the FDA to treat this disease. Although three vaccines have been approved by the FDA, mutations in the SARS-CoV-2 may cause problems in antibody neutralization against the virus. COVID-19 patients have been found either symptomatic or asymptomatic. In most people, the disease was found with mild symptoms with no need for hospitalization, or sometimes patients don't show any symptom. Elderly people and people with compromised health are mainly affected by the disease. Serologic assays involving IgM and IgG antibodies to detect antibodies against SARS-CoV-2 are of great interest as these antibodies can be detected from the second week of the start of COVID-19 symptom's where IgM can be detected after the fourth day of infection and IgG has been found after the eighth day of disease onset. Serologic assays provide quick diagnostic by avoiding PCR false positive/false negative result as well as these provide antibody pattern for estimation of strength and duration of humoral immunity. Here, serologic assays will be used to estimate IgM and IgG antibodies in symptomatic or asymptomatic COVID subjects recovered from the disease.

DETAILED DESCRIPTION:
SARS-CoV-2 (Severe Acute Respiratory Syndrome Coronavirus 2) pandemic has affected millions of people around the globe. Despite many efforts to find some effective medicines against SARS CoV-2, still no established therapeutics available. A year ago, SARS-CoV-2 emerged as a novel virus with no available treatment option and caused a serious disaster across the world. The disease caused by this virus, "COVID-19", announced a global pandemic on March 11, 2020. Without any proper treatment and vaccine for COVID-19, people around the world are currently experiencing a worldwide emergency affecting all societies, and it has sent billions of people into lockdown. Around the world, desperate efforts are underway to curtail this pandemic while it has resulted in the collapsing of health systems and has triggered lasting geopolitical and economic changes. To date, no approved medical treatment is available, which makes social distancing the only best possible solution to stop the spread of the virus. It is thought that future outbreaks of CoVs are unavoidable because of changes in the climate and ecology and increased interaction of humans with animals. Therefore, there is a need to develop effective therapeutics and vaccines against CoVs.

Poor diagnosis of COVID-19 has also contributed to disease severity due to stress (in case of false positive) and disease spread (in case of a false negative). A lack of RT-PCR test sampling of lower tract respiratory specimens was the main reason for the misclassification of symptomatic patients as either having COVID-19 or not. A prompt diagnosis with serological testing shows SARS-CoV-2 IgG/IgM patterns in a better and understandable way of seroconversion.

The IgG/IgM assays to detect the length and origin of humoral responses against SARS-CoV-2 is very important, and these antibodies can be detected from a few days after the onset of diseases and may remain in the body even after years of infection. In the case of COVID-19, IgM and IgG response can be observed from the second week of the disease.

In Coronaviruses, IgM and IgG levels are found to disappear over time in humans. IgG antibodies against SARS-CoV-1 were found to wane approximately two years after infection, and the person may become vulnerable to reinfection after the complete reduction of the immune response. In MERS- CoV, IgG levels were found gradually reduced after a year of infection onset. The length of the protective immunity is very important to avoid reinfection and also helps in the prediction of vaccine response in the body. The humoral immune response varies among young and elderly people, men and women, healthy and health compromised people. Studies on dynamics and the mechanisms of the humoral immune response may help in COVID-19 vaccine development and laws implementation, and other public health responses. This study is particularly designed to access the IgM and IgG antibodies in various COVID-19 subjects in Sargodha, Punjab, Pakistan, where no specific study of this kind has been performed. This will help predict the reinfection probabilities among the local population and predict the length and efficacy of the vaccine and the requirement of vaccine boosters.

ELIGIBILITY:
Inclusion Criteria:

* Suspected/PCR positive COVID-19 patients
* Patients aged >18 years and < 60 year
* Able to fill/understand/answer the questionnaire and provide consent to use of personal health information.

Exclusion Criteria:

* Impaired/disable patients who can not understand or provide questionnaire answers
* Patients aged <18 years and > 60 year

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Local people living in the Sargodha District
Sampling Method: Probability Sample
Enrollment: 373 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
IgG positive | from date of consent to date of test completion, up to 40 days
  COVID patients

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Fayyaz U Rehman, PhD, Principal Investigator — University of Sargodha
Locations (2):
- Pakistan (2):
  - University of Sargodha, Sub campus Bhakkar, Bhakkar, Punjab Province
  - University of Sargodha, Sargodha, Punjab Province

REFERENCES:
- [Background] Rehman MFU, Fariha C, Anwar A, Shahzad N, Ahmad M, Mukhtar S, Farhan Ul Haque M. Novel coronavirus disease (COVID-19) pandemic: A recent mini review. Comput Struct Biotechnol J. 2021;19:612-623. doi: 10.1016/j.csbj.2020.12.033. Epub 2020 Dec 31. PMID 33398233
- [Background] Lee YL, Liao CH, Liu PY, Cheng CY, Chung MY, Liu CE, Chang SY, Hsueh PR. Dynamics of anti-SARS-Cov-2 IgM and IgG antibodies among COVID-19 patients. J Infect. 2020 Aug;81(2):e55-e58. doi: 10.1016/j.jinf.2020.04.019. Epub 2020 Apr 23. No abstract available. PMID 32335168